CLINICAL TRIAL: NCT05596448
Title: Investigation of the Efficiency of Coccygeal Nerve Radiofrequency Treatment in Coccydynia'
Brief Title: Coccygeal Nerve Radiofrequency Treatment in Coccydynia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Principal Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Coccygeal Nerve
Record Dates: First submitted 2022-10-22; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Coccyx Disorder
Keywords: coccydinia; coccygeal nerve; radiofrequency ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cocygeal nerve radiofrequency ablation group (Active Comparator): During the procedure, after imaging the sacral and coccygeal corns with ultrasonography, a radiofrequency ablation needle is inserted at the level of the coccygeal horn and radiofrequency ablation is applied at 90 degrees for 60 seconds.
  Interventions: Procedure: Coccygeal nerve radiofrequency ablation
- Conservative treatment group (No Intervention): This group includes patients receiving conservative treatment such as nonsteroidal anti-inflammatory group drugs, physical therapy, and exercise for coccygeal pain.

INTERVENTIONS:
Procedure: Coccygeal nerve radiofrequency ablation — During the procedure, after imaging the sacral and coccygeal corns with ultrasonography, a radiofrequency ablation needle is inserted at the level of the coccygeal horn and radiofrequency ablation is applied at 90 degrees for 60 seconds.
  Arms: Cocygeal nerve radiofrequency ablation group

SUMMARY:
Coccydynia or coccygeal pain is a painful syndrome that affects the coccyx region. The most important etiological factors in the formation of coccidynia are; external and internal trauma. Patients with coccydynia typically complain of coccyx pain. This pain increases with prolonged sitting, bending backwards during sitting, standing for long periods of time, and standing up after sitting. Conservative treatments such as nonsteroidal anti-inflammatory drugs (NSAIDs), levator sudden relaxation exercises, seat cushions, and transcutaneous electrical simulation have all been used to relieve pain, but these methods are ineffective in 10% of patients. In the patient group unresponsive to conservative treatments, there are various interventional treatment options, including caudal epidural steroid injection, ganglion impar blocks, radiofrequency ablation of the sacral nerves, block of the coccygeal nerves and radiofrequency ablation, and coccygectomy.

DETAILED DESCRIPTION:
In algoloji clinic, routinely apply ultrasound-guided coccygeal nerve block and radiofrequency ablation to patients with coccydynia. During the procedure, after imaging the sacral and coccygeal corns with ultrasonography, a radiofrequency ablation needle is inserted at the level of the coccygeal horn and radiofrequency ablation is applied at 90 degrees for 60 seconds. Patients are followed for a while in our post-procedure service for possible hypotension and allergic reactions. In this study, it was planned to apply the Visual Pain Scale (VAS) and Paris Functional Coccydynia Questionnaire at the 1st week, 1st month and 3rd months after the treatment to patients who had coccygeal nerve block and radiofrequency ablation in our clinic due to the complaint of coccydynia resistant to conservative treatment methods. In this way, it is planned to evaluate the efficacy of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Coccygeal pain

Exclusion Criteria:

* Malignancy
* İnfection
* Coagulation disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-22 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Paris Functional Coccydynia Questionnaire | 4 weeks
  It is a scale that measures the severity of coccygeal pain. Scored between ''0: no pain'' and ''10: worst pain.

SECONDARY OUTCOMES:
Visual analog scale (VAS) | 4 weeks
  It is a scale that measures the severity of pain. In this questionnaire, the patient's pain in sitting position, getting up from sitting position, standing and walking, traveling and at night is recorded. Scored between ''0: no pain'' and ''10: worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Taylan Akkaya, Study Director — Diskapi Yildirim Beyazıt Teaching and Research Hospital; Gevher Rabia Genç Perdecioğlu, Study Chair — Diskapi Yildirim Beyazıt Teaching and Research Hospital; Hüseyin Alp Alptekin, Study Chair — Diskapi Yildirim Beyazıt Teaching and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazıt Teaching and Research Hospital, Ankara, Turkey (Türkiye)